CLINICAL TRIAL: NCT07190001
Title: An Exploratory Clinical Study to Evaluate the Safety and Efficacy of YOLT-204 in Patients With Hemoglobinopathies (β-thalassemia and Sickle-cell Disease)
Brief Title: YOLT-204 in Patients With Hemoglobinopathies
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Guangzhou Women and Children's Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YOLT-204-IIT-002
Record Dates: First submitted 2025-09-16; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Hemoglobinopathies (Transfusion-dependent β-thalassemia and Sickle Cell Disease)
MeSH Terms: conditions — Hemoglobinopathies; Anemia, Sickle Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arms (Experimental): The intervention group will receive YOLT-204 on day0
  Interventions: Drug: YOLT-204

INTERVENTIONS:
Drug: YOLT-204 — The intervention group will receive YOLT-204 on day0

SUMMARY:
This is a single-arm, open-label, single-dose, dose-escalation trial that plans to enrol 3-18 patients with transfusion-dependent β-thalassaemia (TDT) or sickle-cell disease (SCD). Its primary aims are to evaluate the safety and tolerability of a single administration of YOLT-204 and to obtain preliminary data on its effect on plasma fetal-haemoglobin levels. The main-study screening period may last up to 60 days; the treatment day is Day 0 (D0). Safety follow-up continues through Week 52 post-dose. After completion of the main study, participants will enter long-term follow-up extending to 15 years post-dose.

ELIGIBILITY:
Inclusion Criteria:

* Aged 3-17 years (inclusive); any sex.
* The subject and/or his/her legally authorized guardian/representative must fully understand the study and voluntarily sign a written informed-consent form.
* Karnofsky Performance Status (KPS) ≥ 70 (if ≥ 16 years old) or Lansky Performance Scale (LPS) ≥ 70 (if < 16 years old).
* Detailed medical records of red-cell transfusions during the 2 years before informed-consent signature must be available, including volume or units transfused and pre-/post-transfusion red-cell and hemoglobin levels.
* No severe hematopoietic dysfunction; cardiac, pulmonary, hepatic, and renal function essentially normal.
* Coagulation: international normalized ratio (INR) and activated partial thromboplastin time (APTT) ≤ 1.5 × upper limit of normal (ULN).
* Renal function: serum creatinine ≤ 1.5 × ULN; if creatinine > 1.5 × ULN, calculated creatinine clearance > 50 mL/min by the Schwartz formula.
* Hepatic function: alanine aminotransferase (ALT) ≤ 3 × ULN and aspartate aminotransferase (AST) ≤ 3 × ULN.
* Cardiac function: left-ventricular ejection fraction (LVEF) ≥ 50 %.
* Good compliance; willing to adhere to visit schedules, study procedures, laboratory tests, and other protocol requirements.
* Agrees to use at least one highly effective contraceptive method from informed-consent signature through the end of the main study (Week 52 visit).
* Willing to participate in long-term follow-up.
* Screening genotype shows HbSS or HbSβ0; prior reports acceptable if assessed as adequate by the investigator.
* If on L-glutamine, regimen must have been stable for ≥ 3 months before study-drug administration; if on hydroxyurea, must have discontinued ≥ 8 weeks before study-drug administration.
* Meets severe SCD criteria: despite optimal supportive therapy (including, but not limited to, analgesics and hydroxyurea), at least two of the following events occurred in the 12 months before screening:
* Severe intermittent acute pain requiring healthcare-provider management;
* Acute chest syndrome with new pulmonary infiltrate on chest imaging plus pneumonia-like symptoms, pain, or fever;
* Splenic sequestration crisis manifested by enlarged spleen, left upper-quadrant pain, and acute Hb drop > 20 g/L.

Exclusion Criteria:

* 1.History of multiple drug allergies or hypersensitivity to oligonucleotides or lipid nanoparticles (LNP).

  2.Clinically significant active bacterial, viral, fungal, or parasitic infection at screening, as judged by the investigator.

  3.White blood cell (WBC) count < 3 × 10⁹/L and/or platelet count < 100 × 10⁹/L at screening.

  4.Uncorrected bleeding diathesis. 5.Massive splenomegaly at screening (spleen edge below the umbilicus or > 4 cm below the costal margin) deemed by the investigator to preclude enrollment.

  6.Serum ferritin ≥ 5 000 ng/mL, or MRI T2* evidence of severe cardiac or hepatic iron overload.

  7.Positive for hepatitis B surface antigen (HBsAg), anti-hepatitis C virus antibody, anti-HIV antibody, or specific anti-Treponema pallidum antibody.

  8.Prior hematopoietic stem-cell transplantation, gene therapy, or gene-editing therapy.

  9.Participation in another clinical trial and receipt of investigational product within 3 months before first dose of study drug.

  10.Current or prior malignancy, myeloproliferative disorder, or immunodeficiency disease.

  11.Severe psychiatric illness precluding cooperation; clinically significant pulmonary hypertension requiring medical intervention; recent malaria; first-degree relative with hematologic malignancy.

  12.Positive pregnancy test, pregnancy, or lactation in female subjects at screening.

  13.Any condition (past or present) that, in the investigator's opinion, could confound results, compromise participation, or render the patient unsuitable for the study.

  14.Use within 3 months before study drug: erythropoietin (EPO), thalidomide, hydroxyurea, luspatercept, or similar agents.

  15.In subjects ≥ 12 years, abnormal transcranial Doppler (TCD) with middle cerebral or internal carotid artery velocity ≥ 200 cm/s.

  16.History of moyamoya disease or imaging findings consistent with moyamoya at screening, assessed by the investigator as conferring bleeding risk.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Adverse event rate | From baseline to 52 weeks after dose
  Calculate the rate of various adverse events
3 months of sustained transfusion reduction | From baseline to 52 weeks after dose
  Analysis begins one month after treatment with YOLT-204, and the proportion of patients who achieve at least 3 months of sustained transfusion reduction (sustained TR3) is obtained.
3 months of sustained HbF level ≥20% | From baseline to 52 weeks after dose
  Proportion of patients who, starting one month after YOLT-204 treatment and without concomitant hydroxyurea, maintain HbF ≥ 20 % for at least three consecutive months.

SECONDARY OUTCOMES:
The proportion of alleles with intended modifications | From baseline to 52 weeks after dose
  The proportion of alleles with intended modifications in peripheral blood leukocytes and bone marrow cells
Concentration of Hemoglobin | From baseline to 52 weeks after dose
  The concentration of Hemoglobin was measured by laboratory
Concentration of Fetal hemoglobin | From baseline to 52 weeks after dose
  The concentration of Fetal hemoglobin was measured by laboratory
Concentration of proportion of F cell | From baseline to 52 weeks after dose
  The proportion of F cell was measured by laboratory
3 months of transfusion independence | From baseline to 52 weeks after dose
  Analysis begins one month after treatment with YOLT-204, and the proportion of patients who achieve at least 3 months of transfusion independence (sustained TI3) is obtained.
6 months of sustained transfusion reduction | From baseline to 52 weeks after dose
  Analysis begins one month after treatment with YOLT-204, and the proportion of patients who achieve at least 6 months of sustained transfusion reduction (sustained TR6) is obtained.
6 months of transfusion independence | From baseline to 52 weeks after dose
  Analysis begins one month after treatment with YOLT-204, and the proportion of patients who achieve at least 6 months of transfusion independence (sustained TI6) is obtained.
Free of hospitalization due to vaso-occlusive crisis | From baseline to 52 weeks after dose
  Analysis begins one month after treatment with YOLT-204, and the proportion of patients who remained free of hospitalization due to vaso-occlusive crisis.
Free of any vaso-occlusive crisis | From baseline to 52 weeks after dose
  Analysis begins one month after treatment with YOLT-204, and the proportion of patients who remained free of any vaso-occlusive crisis
Change of red-blood-cell transfusions given | From baseline to 52 weeks after dose
  Analysis begins one month after treatment with YOLT-204, and the Change from baseline in volume of red-blood-cell transfusions given for SCD-related indications
The number of vaso-occlusive crises | From baseline to 52 weeks after dose
  Change from baseline in the number of vaso-occlusive crises within 1 year after YOLT-204 treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou women and children's medical center, Guangzhou, Guangdong, China